CLINICAL TRIAL: NCT02342938
Title: Simultaneous MEG or fMRI And INtracranial EEG
Acronym: SEMAINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: University of Konstanz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011.698
Record Dates: First submitted 2014-10-06; First posted 2015-01-21 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; Healthy Volunteers
Keywords: Epilepsy surgery; High frequency activity; icEEG; fMRI; MEG
MeSH Terms: conditions — Epilepsy | interventions — Magnetoencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient (Experimental)
  Interventions: Procedure: fMRI
- Volunteers (Experimental)
  Interventions: Procedure: MEG or fMRI And INtracranial EEG

INTERVENTIONS:
Procedure: MEG or fMRI And INtracranial EEG
  Arms: Volunteers
Procedure: fMRI
  Arms: Patient

SUMMARY:
The SEMAINE project will investigate intracranial EEG (icEEG) simultaneously recorded with either fMRI or MEG to 1) improve identification of the epileptogenic zone in patients suffering from drug-resistant partial epilepsy, and 2) define the functional organization of neural networks underlying human perception and cognition in order to prevent inadvertent deficits resulting from neurosurgical resection. In particular, high-frequency activity (HFA), as measured with icEEG, has been demonstrated in recent years as a relevant index for both epileptogenic tissue and healthy cortical processing, but its correlates in fMRI and MEG require further investigation. This will be a pioneering effort in several respects, as the first to directly measure high-frequency neural activity in tandem with fMRI, and among the first to do so with MEG. In addition to their attractiveness as noninvasive imaging techniques, fMRI and MEG have the potential to examine whole-brain networks that are not accessible to icEEG's necessarily limited spatial coverage. Furthermore, such a campaign of simultaneous recordings will take unprecedented advantage of icEEG as the bridge between the two noninvasive techniques, providing compelling evidence for the links between all three measurements with respect to underlying high-frequency neural activity in both health and disease. This project will therefore lead to improved selection of epilepsy surgery candidates and improved neurosurgical outcomes from the precise mapping of epileptogenic and healthy brain networks. The same techniques will be immediately applicable to functional mapping of other types of neurosurgery populations as well as diagnostic neuroimaging of neurological and psychiatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 60 years, not subject of any measure of legal protection
* Patients suffering from drug resistant partial epilepsy
* Patient undergoing intracranial video EEG
* Patients with electrodes implanted in orthogonal
* no MRI cons-indication
* Patients who signed a consent form
* Intellectual capacity to perform cognitive tasks and to sign an informed consent.
* Affiliation to social security

Exclusion Criteria:

* Pregnant women
* Elderly patients under 18 or over 60 years Patient not suffering from drug resistant partial epilepsy, or not scheduled for a SEEG
* MRI cons-indication
* Patients taking psychotropics drugs
* Claustrophobia
* Inability to perform cognitive tasks or to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Blood Oxygenation Level Dependent changes, associated with intracranial EEG signal, as determined by simultaneous fMRI and icEEG | Month 2
  fMRI correlates of epileptic and cognitive-induced high-frequency activities
MEG signal, associated with intracranial EEG signal, as determined by simultaneous MEG and icEEG | Month 2
  MEG correlates of epileptic and cognitive-induced high-frequency activities

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Background] Saignavongs M, Ciumas C, Petton M, Bouet R, Boulogne S, Rheims S, Carmichael DW, Lachaux JP, Ryvlin P. Neural Activity Elicited by a Cognitive Task can be Detected in Single-Trials with Simultaneous Intracerebral EEG-fMRI Recordings. Int J Neural Syst. 2017 Feb;27(1):1750001. doi: 10.1142/S0129065717500010. Epub 2016 Aug 22. PMID 27718767